CLINICAL TRIAL: NCT05068466
Title: A Phase 1, Double-Blind, Randomized, Placebo-Controlled, Multiple Dose-Escalation Study to Assess the Safety, Tolerability, and Pharmacokinetics of INCB054707 When Administered Orally to Healthy Japanese Participants
Brief Title: A Study to Evaluate the Safety, Tolerability and Pharmacokinetics of INCB054707
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incyte Biosciences Japan GK (Industry)
Responsible Party: Sponsor
Organization: Incyte Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: INCB 54707-108
Record Dates: First submitted 2021-09-27; First posted 2021-10-05 (Actual); Last update posted 2022-09-16 (Actual); Status verified 2022-09

CONDITIONS: Healthy Participants
Keywords: INCB054707

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- INCB054707 (Dose A) (Experimental): Participants will be administered single-dose INCB054707 on Day 1 followed by once daily dose of INCB054707 on Days 5 to 12 (8 doses) administered orally after a fast of ≥ 8 hours
  Interventions: Drug: INCB054707
- INCB054707 (Dose B) (Experimental): Participants will be administered a single-dose INCB054707 on Day 1 followed by once daily dose of INCB54707 on Days 5 to 12 (8 doses) administered orally after a fast of ≥ 8 hours.
  Interventions: Drug: INCB054707
- Placebo (Dose A) (Placebo Comparator): Participants will be administered single-dose placebo on Day 1 followed by once daily dose of placebo on Days 5 to 12 (8 doses) administered orally after a fast of ≥ 8 hours
  Interventions: Drug: Placebo
- Placebo (Dose B) (Placebo Comparator): Participants will be administered single-dose placebo on Day 1 followed by once daily dose of placebo on Days 5 to 12 (8 doses) administered orally after a fast of ≥ 8 hours
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: INCB054707 — Administered Orally
  Other Names: Povorcitinib
  Arms: INCB054707 (Dose A); INCB054707 (Dose B)
Drug: Placebo — Administered Orally
  Arms: Placebo (Dose A); Placebo (Dose B)

SUMMARY:
This is a single-center, randomized, double-blind, placebo-controlled, sponsor-unblinded, Phase 1 study designed to evaluate the safety, tolerability, and PK of escalating oral doses of INCB054707 in healthy male Japanese participants. Participants in each cohort will be divided into placebo or INCB054707 by a 3:1 INCB054707:placebo random assignment.

ELIGIBILITY:
Inclusion Criteria:

* Male healthy Japanese adult participants aged 20 to 55 years with a minimum weight of 48 kg.
* Body mass index between 18.0 and 30.5 kg/m2.
* No clinically significant findings in screening evaluations.
* Ability to swallow and retain oral medication.
* Willingness to avoid fathering children

Exclusion Criteria:

* History of clinically significant cardiovascular, respiratory, renal, gastrointestinal, endocrine, hematopoietic, psychiatric, and/or neurological disease.
* History of rheumatologic/autoimmune disorders, except for minor eczema and rosacea.
* Resting pulse < 40 bpm or > 100 bpm, confirmed by repeat testing at screening.
* History or presence of an abnormal ECG before initial dose administration that, in the investigator's opinion, is clinically significant.
* Presence of a malabsorption syndrome possibly affecting drug absorption (eg, Crohn's disease or chronic pancreatitis).
* Hemoglobin, WBC, platelet, or ANC that is out of the laboratory's range unless considered clinically insignificant by the investigator at screening or check-in.
* History of malignancy within 5 years of screening, with the exception of cured basal cell or squamous cell carcinoma of the skin.
* Current or recent (within 6 months of screening) clinically significant gastrointestinal disease or surgery (including cholecystectomy, excluding appendectomy) that could affect the absorption of study drug.
* Any major surgery within 6 months of screening.
* Donation of blood to a blood bank or in a clinical study (except a screening visit) within 4 weeks of screening (within 2 weeks for plasma donation).
* Blood transfusion within 4 weeks of check-in.
* Chronic or current active infectious disease requiring systemic antibiotic, antifungal, or antiviral treatment
* Positive test for HIV and known active HBV or HCV infection or risk of reactivation of HBV or HCV.
* History of alcoholism within 3 months of screening.
* Positive breath or urine test for ethanol or positive urine screen for drugs of abuse that are not otherwise explained by permitted concomitant medications or diet.
* Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) before the first dose of study drug with another investigational medication or current enrollment in another investigational drug study.
* Current treatment or treatment within 30 days or 5 half-lives (whichever is longer) before the first dose of study drug with an inducer or inhibitor of CYP3A4, P-gp, or BCRP
* Current use of prohibited medication
* Consumption of Seville oranges, grapefruit or grapefruit juice, pomelos, exotic citrus fruits, grapefruit hybrids, or fruit juices within 72 hours before the first dose of study drug.
* History of any significant drug allergy (such as anaphylaxis or hepatotoxicity) deemed clinically relevant by the investigator.
* Known hypersensitivity or severe reaction to INCB054707 or any excipients of INCB054707
* Inability to undergo venipuncture or tolerate venous access.
* Inability or unlikeliness of the participant to comply with the dose schedule and study evaluations, in the opinion of the investigator.
* History of tobacco- or nicotine-containing product use within 1 month of screening.
* Use of prescription drugs within 14 days of study drug administration or nonprescription medications/products within 7 days of study drug administration.
* Any condition that would, in the investigator's judgment, interfere with full participation in the study.
* Positive syphilis test.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 30 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2022-01-25 (Actual); Study Completion 2022-01-25 (Actual)

PRIMARY OUTCOMES:
Number of participants with Treatment Emergent Adverse Events (TEAE'S) | 3 months
  Adverse events reported for the first time or worsening of a pre-existing event after first dose of study drug/treatment.
Pharmacokinetics Parameter : Cmax of INCB054707 | 17 Days
  Maximum Observed Plasma Concentration of INCB054707
Pharmacokinetics Parameter : Cmin of INCB054707 | 17 Days
  Minimum Observed Plasma Concentration of INCB054707
Pharmacokinetics Parameter : tmax of INCB054707 | 17 Days
  Time to reach maximum plasma concentration of INCB054707
Pharmacokinetics Parameter : AUC(0-t) of INCB054707 | 17 Days
  Area Under the concentration- time curve up to the last measurable concentration of INCB054707
Pharmacokinetics Parameter : AUC(0-∞) of INCB054707 | 17 Days
  Area Under the Concentration-time Curve From 0 to Infinity of INCB054707
Pharmacokinetics Parameter : AUC(0-tau) of INCB054707 | 17 Days
  Area under the single-dose or steady-state plasma concentration-time curve from hour 0 to the end of the dosing period of INCB054707

SECONDARY OUTCOMES:
Pharmacokinetics Parameter : t1/2 of INCB054707 | 17 Days
  Pharmacokinetics Parameter : t1/2 of Apparent terminal phase disposition half-life of
Pharmacokinetics Parameter : CL/F of INCB054707 | 17 Days
  Oral dose clearance of INCB054707
Pharmacokinetics Parameter : Vz/F of INCB054707 | 17 Days
  Apparent oral dose volume of distribution of INCB54707
Pharmacokinetics Parameter : Cavg of INCB054707 | 17 Days
  Average plasma concentration at steady state of INCB054707
Pharmacokinetics Parameter : λz of INCB054707 | 17 Days
  Apparent terminal-phase disposition rate constant of INCB054707

CONTACTS AND LOCATIONS:
Locations (1):
- Souseikai Fukuoka Mirai Hospital, Fukuoka, Japan

IPD SHARING:
Plan to Share IPD: Yes
Incyte shares data with qualified external researchers after a research proposal is submitted. These requests are reviewed and approved by a review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  The trial data availability is according to the criteria and process described on https://www.incyte.com/our-company/compliance-and-transparency
Supporting Information: Study Protocol, SAP
Time Frame: Data will be shared after the primary publication or 2 years after the study has ended for market authorized products and indications.
Access Criteria: Data from eligible studies will be shared with qualified researchers according to the criteria and process described in the Data Sharing section of the www.incyteclinicaltrials.com website. For approved requests, the researchers will be granted access to anonymized data under the terms of a data sharing agreement.
URL: https://www.incyte.com/our-company/compliance-and-transparency